CLINICAL TRIAL: NCT00120562
Title: A Gene Expression and Metabolic Profile of Weight Loss: Studies of Patients Following Gastric Bypass Surgery
Brief Title: Studies of Biological Changes Related to Weight Loss After Gastric Bypass Surgery
Status: Terminated | Type: Observational
Sponsor: Rockefeller University (Other)
Collaborators: New York Obesity and Nutrition Research Center (Other)
Other Study IDs: JFN 0385
Record Dates: First submitted 2005-07-11; First posted 2005-07-18 (Estimated); Last update posted 2009-08-28 (Estimated); Status verified 2009-08

CONDITIONS: Obesity; Morbid Obesity; Weight Loss
Keywords: weight loss surgery; gastric bypass surgery
MeSH Terms: conditions — Obesity; Obesity, Morbid; Weight Loss

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Gastric Bypass Surgery

SUMMARY:
Weight loss achieved by dieting induces multiple changes. These changes include a decrease in metabolic rate (the rate in which the body burns its calories), an increase in appetite and other physiological and hormonal changes that may be the cause of failure in dieting. Many of these parameters that have never been evaluated when weight is lost after gastric bypass surgery will be tested in this study.

DETAILED DESCRIPTION:
While gastric bypass surgery (GBS) is known to be highly effective in achieving significant weight loss, it is also associated with other biologic changes that occur in the body when weight is lost. In this study, subjects undergoing gastric bypass surgery will be followed throughout the weight loss period. They will undergo four detailed medical evaluations to assess changes in several biological systems that occur in the body when weight is lost.

The initial assessment will be performed before the surgery (testing period 1). After surgery is completed, subjects will attend clinic visits at the Rockefeller University outpatient clinic. During these visits, weight and leptin levels will be monitored. Two additional assessments will be performed during weight loss, when subjects lose 10% and 20% of their initial weight (testing periods 2 and 3 respectively). A final evaluation will be performed after weight is stabilized, about 18 months after the surgery is completed (testing period 4). Each testing period will be performed over a 2 week period in an inpatient setting at the Rockefeller University Hospital. During testing periods subjects will undergo a series of metabolic, behavioral, hormonal, immune and molecular tests to evaluate changes that occur in the body after weight loss. Subjects will receive monetary compensation for participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years old
* Subjects approved for gastric bypass surgery

Exclusion Criteria:

* Subjects not approved for gastric bypass surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * 18 - 65 years old
  * Subjects approved for gastric bypass surgery
Sampling Method: Probability Sample
Enrollment: 13 (Estimated)
Dates: Start 2007-07

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M. Friedman, MD, Principal Investigator — Rockefeller University
Locations (1):
- St. Luke's Obesity Research Center, NY NY 10023 and New York Hospital, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.rucares.org